CLINICAL TRIAL: NCT05375097
Title: Real-world Impact of Erenumab on Sick-leaves, Health Care Resource Use and Comorbidities Based on Occupational Health Care Registry in Finland: an Observational Retrospective Mirror-image Study (REFI)
Brief Title: Real-world Impact of Erenumab on Sick-leaves, Health Care Resource Use and Comorbidities.
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CAMG334AFI03
Record Dates: First submitted 2022-05-10; First posted 2022-05-16 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Migraine
Keywords: Erenumab,; CGRP,; real world evidence,; sick leaves,; working impairment,; health care visits,; prescriptions,; migraine
MeSH Terms: conditions — Migraine Disorders | interventions — erenumab

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Erenumab responder patients: Patients who met the responder definition of two or more erenumab prescriptions with no evidence of switch to other CGRPi were included in the main analyses
  Interventions: Other: Erenumab
- Migraine controls: Age and gender matched migraine patients on triptan medication, excluding those on botulinum toxin, erenumab and fremanezumab to benchmark the level of HCRU, sick leaves, and medication patterns

INTERVENTIONS:
Other: Erenumab — Patients who met the responder definition of two or more erenumab prescriptions with no evidence of switch to other CGRPi were included in the main analyses
  Groups: Erenumab responder patients

SUMMARY:
This was a retrospective registry-based study utilizing data collected in association with clinical care of patients. All data was stored in electronic health records at Terveystalo data base, and no patients were contacted for the study.

DETAILED DESCRIPTION:
Patients initiating erenumab treatment between 20.9.2018 - 15.10. 2019, and data on sick leave days, diagnoses and health care visits as well as medications based on prescriptions were assessed.

Following time frames for analyses of sick leaves and health care utilization in patients on erenumab treatment and in controls were reported:

Follow-up analyses: For cases (erenumab) with occupational healthcare, a minimum of 12 months on erenumab treatment was required for the analysis of sick leaves and visits

Pre erenumab: Follow-up data before index (defined as the first reimbursement decision/prescription for erenumab, or initiation of erenumab injections (before reimbursement approval)) from the Terveystalo database of those with consent

Post erenumab: Follow-up data after index, from the Terveystalo database of those with consent

Time frames for comparison (sick leaves and visits): One year before index vs. >12 months erenumab after index, One year before index vs. 6-12 months of erenumab after index (patient years), sensitivity analysis

Time frames for comparison (medications): 12 months before index vs. 12 months post follow-up

Controls (triptan treated migraine patients): Corresponding time frames as in cases.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients on erenumab treatment ATC: N02CX07
* Diagnosis of migraine (ICD G43)
* Consented
* Occupational healthcare

Exclusion Criteria:

None

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients on erenumab treatment
Sampling Method: Non-Probability Sample
Enrollment: 162 (Actual)
Dates: Start 2020-07-03 (Actual); Primary Completion 2021-05-14 (Actual); Study Completion 2021-05-14 (Actual)

PRIMARY OUTCOMES:
Number of sick leave days (headache) | throughout the study, approximately 2 years
  Sick leaves included migraine or head-ache related registered sick leave days at Terveystalo in the occupational healthcare cohort and controls.

SECONDARY OUTCOMES:
Change in number of sick leave days (all cause) | throughout the study, approximately 2 years
  Sick leaves included all registered sick leave days at Terveystalo in the occupational healthcare cohort and controls.
Change in number of healthcare visits (head-ache related) | throughout the study, approximately 2 years
  Number of headache related healthcare visits were reported.
Change in number of healthcare visits (all cause) | throughout the study, approximately 2 years
  Number of healthcare visits were reported.
Medication patterns: Number of patients receiving medications of interest | throughout the study, approximately 2 years
  The number of patients receiving medications of interest in erenumab treated patients in migraine patient controls were reported.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, East Hanover, New Jersey, United States

REFERENCES:
- See also: Results for CAMG334AFI03 from the Novartis Clinical Trials Results Database — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17935